CLINICAL TRIAL: NCT04615676
Title: Prospective Evaluation of the Predictive Criteria of Severity Related to Patient Calling Emergency Centre for Low or High Respiratory Infection With or Without Fever and Suspected to be COVID-19.
Brief Title: Prospective Evaluation of the Predictive Criteria of Severity for Respiratory Infection Due to COVID-19 Virus
Acronym: COPREG
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/20/0141
Record Dates: First submitted 2020-11-03; First posted 2020-11-04 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: SARS-CoV2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Follow-up phone call — Follow-up phone call after month to detect which patient have been hospitalized

SUMMARY:
Emergency call centers are very solicited in epidemic situations. It is necessary to detect early Predictive Criteria of Severity in COVID respiratory infection to identify patients at risk of complication or aggravation from an emergency call center in order to adapt their orientation and their medical management.

ELIGIBILITY:
Inclusion Criteria:

* patient (more than 15 years old) calling the emergency call center (15 center) for Low or High Respiratory Infection With or Without Fever and Suspected to be COVID

Exclusion Criteria:

* unknown contact facility
* call not regulated by a practitioner from the medical emergency help team

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patient (more than 15 years old) calling the emergency call center (15 center) for Low or High Respiratory Infection With or Without Fever and Suspected
Sampling Method: Probability Sample
Enrollment: 4734 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2020-07-17 (Actual)

PRIMARY OUTCOMES:
Hospitalization | Month 1
  Hospitalization declared by the patient 1 month after his call to the emergency call center

CONTACTS AND LOCATIONS:
Overall Officials: Charles-Henri HOUZE-CERFON, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided